CLINICAL TRIAL: NCT00831285
Title: A Double-Blind, Randomized, Controlled Study to Examine the Glycemic Response of Barley Tortillas in Healthy Volunteers
Brief Title: Barley Tortillas Study in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Dr. Carla Taylor, Department of Human Nutritional Science, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: B2008:133; Agriculture and Agri-food CAN
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- tortilla with high amylose flour (Experimental)
  Interventions: Dietary Supplement: food product
- barley tortilla with low amylose flour (Experimental)
  Interventions: Dietary Supplement: food product
- barley tortilla with low amylose flour and soluble fibre (Experimental)
  Interventions: Dietary Supplement: food product
- barley tortilla with low amylose flour and insoluble fibre (Experimental)
  Interventions: Dietary Supplement: food product
- glucose (Active Comparator)
  Interventions: Dietary Supplement: food product
- barley tortilla with low amylose flour and low soluble fibre (Experimental)
  Interventions: Dietary Supplement: food product

INTERVENTIONS:
Dietary Supplement: food product — food product given at one of six visits

SUMMARY:
The variation in starch and fibre composition of prepared barley tortillas will have a significant effect on glycemic response.

DETAILED DESCRIPTION:
Specifically, we wish to examine the glycemic response of barley tortillas containing different ratios of amylose and amylopectin and different amounts of soluble and insoluble fibre with an appropriate control during acute phase testing in healthy volunteers. Possible relationships between composition of the barley tortillas and the degree of physiological response will also be investigated as the secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* male or female age 18 to 40 years
* normal glycated hemoglobin of <6%
* BMI of 20 to 30
* must read the consent form
* must comply with the protocol requirements

Exclusion Criteria:

* allergies to barley flour
* presence of chronic conditions such as cardiovascular disease, hypertension, disorders affecting the gastrointestinal tract, thyroid disease, and requiring medication for these conditions
* requiring medication for glycemic control
* consumption of supplements which have an effect on blood glucose response

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Calculation of area under the curve for glucose and insulin | 6 weeks

SECONDARY OUTCOMES:
comparison of food groups using ANOVA | 6 weeks
measurement of incretins | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface General Hospital Research Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Makelainen H, Anttila H, Sihvonen J, Hietanen RM, Tahvonen R, Salminen E, Mikola M, Sontag-Strohm T. The effect of beta-glucan on the glycemic and insulin index. Eur J Clin Nutr. 2007 Jun;61(6):779-85. doi: 10.1038/sj.ejcn.1602561. Epub 2006 Dec 6. PMID 17151593
- See also: Canadian Centre for AgriFood Research in Health and Medicine — http://www.sbrc.ca/ccarm